CLINICAL TRIAL: NCT03699293
Title: NSAIDs vs. Coxibs in the Presence of Aspirin: Effects on Platelet Function, Endothelial Function, and Biomarkers of Inflammation in Subjects With Rheumatoid Arthritis and Increased Cardiovascular Risk or Cardiovascular Disease
Brief Title: NSAIDs vs. Coxibs in the Presence of Aspirin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-2915
Record Dates: First submitted 2018-09-21; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases | interventions — Celecoxib; Naproxen; Tablets; Aspirin

STUDY DESIGN:
Intervention Model Description: Qualified patients will be treated with immediate release 81mg aspirin for 4 weeks in the run-in period followed by randomization to celecoxib (200 mg bid) vs. naproxen sodium (550 mg bid) for 4 weeks and then cross over to the other drug for another 4 weeks. Blood and urine samples will be collected before the aspirin run-in period (baseline), 24±4 hrs after the last dose of aspirin in the run-in period, 24±4 hr after the last dose of the study drug in the first period and 24±4 hr after the last dose of the study drug in the second period. Assays for platelet function, biomarkers of inflammation and endothelial function will be performed at these time points
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASA and Celecoxib (Active Comparator): Take celecoxib 200mg capsule twice a day and aspirin 81mg tablet once a day for 4 weeks (after completion of the run-in period)
  Interventions: Drug: celecoxib 200mg capsule; Drug: Aspirin 81mg tablet
- ASA and Naproxen (Active Comparator): Take naproxen sodium 550mg tablet twice a day and aspirin 81mg tablet once a day (after completion of the run-in period)
  Interventions: Drug: naproxen sodium 550mg tablet; Drug: Aspirin 81mg tablet

INTERVENTIONS:
Drug: celecoxib 200mg capsule — celecoxib 200mg twice a day for 4 weeks
  Other Names: Celebrex
  Arms: ASA and Celecoxib
Drug: naproxen sodium 550mg tablet — naproxen sodium 550mg twice a day for 4 weeks
  Other Names: Aleve; Naprosyn
  Arms: ASA and Naproxen
Drug: Aspirin 81mg tablet — 81mg aspirin for 4 weeks in the run-in period, and for 8 weeks during treatment and crossover period
  Other Names: Bayer Aspirin

SUMMARY:
The objectives of this single site, randomized, crossover study is to evaluate the pharmacodynamic interactions between aspirin, NSAIDs and Coxibs with respect to platelet function, biomarkers of inflammation and endothelial function.

DETAILED DESCRIPTION:
The relative cardiovascular safety of NSAIDs, particularly among patients with cardiovascular disease (CVD) or at higher CVD risk, has generated considerable concern among both patients and physicians because of knowledge gaps in the evidence relative to comparative safety and pharmacodynamic interactions between aspirin and NSAIDs. In the recently reported PRECISION trial, a moderate dose of celecoxib was found to be noninferior to ibuprofen or naproxen with respect to cardiovascular safety in patients with arthritis at increased CVD risk. At this time, no comparative prior data are available analyzing the effects of NSAIDs vs. Coxibs in the presence of aspirin on platelet function, biomarkers of inflammation and endothelial function.

Thirty patients with rheumatoid arthritis who are at high cardiovascular (CV) risk or with established CV disease will be enrolled in the study. Patients taking anticoagulant therapy or any other antiplatelet agent other than aspirin will be excluded.

Patients will be treated with immediate release 81mg aspirin for 4 weeks in the run-in period followed by randomization to celecoxib (200 mg bid) vs. naproxen sodium (550 mg bid) for 4 weeks and then cross over to the other drug for another 4 weeks. Blood and urine samples will be collected at baseline before the aspirin run in period, 24±4 hr after the last dose of aspirin in the run in period, 24±4 hr after the last dose of the first period study drug and 24±4 hr after the last dose of the second period study drug. Assays for platelet function, biomarkers of inflammation and endothelial function will be performed at these time points.

ELIGIBILITY:
Inclusion Criteria:Qualified patients should have all 4 main criteria

1. Age 18-75 years of age for patients who regularly use NSAIDs.
2. Age 18-65 years of age for patients who do not regularly use NSAIDs
3. Able to give informed consent
4. Subjects with CVD or increased CV risk. Please see definitions for each criteria below:

   * Increased CV risk (Subjects should have at least 3 of the following)

     * > 55 years of age
     * Hypertension
     * Dyslipidemia (LDL > 160 mg/dL or HDL < 40 mg/dL in females and < 35 mg/dL in males or subjects currently receiving lipid lowering therapy as standard of care (i.e. statin drugs, prescription ω 3-acid ethyl esters, fibrates or prescription niacin [≥1,000 mg/d])
     * Family history of premature CV disease (MI, angina pectoris, heart failure, cardiac death or coronary revascularization, stroke, carotid endarterectomy, or other arterial surgery or angioplasty for atherosclerotic vascular disease in a parent, grandparent, or sibling with symptom onset or diagnosis before age 55 y for males and 65 y for females)
     * Current smoker
     * Left ventricular hypertrophy
     * Documented ankle brachial index of <0.9
     * History of microalbuminuria, urine protein-creatinine ratio of >2
   * CV disease (defined as one of the following):

     * Calcium score of >0
     * ≥ 50 % occlusion of a coronary artery by angiography
     * ≥ 50 % occlusion of a carotid artery by angiography or ultrasound
     * History of stable angina
     * Symptomatic peripheral arterial disease
     * Prior MI, unstable angina, percutaneous coronary intervention, CABG, TIA, ischemic stroke, carotid endarterectomy, or other arterial surgery or angioplasty, which have occurred > 3 months prior to screening visit
     * Diabetes Mellitus type 1 or 2 (considered a CV disease equivalent).
   * Clinical diagnosis of rheumatoid arthritis, as determined by individual patient and physician, requiring daily treatment with NSAIDs.

Exclusion Criteria: Subjects with any of the following criteria will be excluded from this study:

1. Unstable angina, MI, CVA, CABG <3 months from screening visit
2. Planned coronary, cerebrovascular, or peripheral revascularization
3. Undergone major surgery within 3 months prior to screening visit or has planned major surgery during the study period
4. Uncontrolled hypertension (SBP >190, DBP >100 mm Hg) during screening visit
5. Uncontrolled arrhythmia < 3 months from screening visit
6. NYHA class III-IV heart failure or if available, ejection fraction ≤ 35 %
7. Within 6 months prior to screening visit, a history of ACS or hospitalization for heart failure
8. Oral corticosteroid, prednisone (or equivalent) > 20 mg daily
9. Anticoagulation therapy
10. Antiplatelet therapy except for aspirin
11. GI ulceration < 60 days before screening visit
12. GI bleeding, perforation, obstruction < 6 months of screening visit
13. Inflammatory bowel disease, diverticulitis active < 6 months of screening visit
14. AST, ALT, or BUN >2x the upper limit normal (within 30 days prior to screening visit)
15. Creatinine level >1.7 mg/dL in men, 1.5 mg/dL in women (within 30 days prior to screening visit)
16. On fluconazole, methotrexate, or lithium therapy
17. Malignancy < 5 years before screening visit
18. Other known, active, significant GI, hepatic, renal, or coagulation disorders
19. Allergy, allergic-type reactions or hypersensitivity (e.g. asthma, urticaria, etc.) to any of the study medications and its components (i.e. sulfonamides)
20. History of any disease of condition that, in the opinion of the investigator would place the subject at an unacceptable risk to participate in this study
21. Any clinically relevant abnormal findings in physical examination, vital signs, or previous laboratory works that, in the opinion of the investigator, may compromise the safety of the subject to participate
22. Subjects who are legally institutionalized
23. Lactating females or females of childbearing potential except for those who are surgically sterile or postmenopausal-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-22 (Actual); Primary Completion 2019-09-24 (Estimated); Study Completion 2019-11-24 (Estimated)

PRIMARY OUTCOMES:
Platelet aggregation | 12 weeks
  Change in platelet aggregation by light transmittance aggregometry between treatment groups

SECONDARY OUTCOMES:
Serum TxB2 | 12 weeks
  Changes in serum TxB2 between treatment groups
Urine thromboxane | 12 weeks
  Changes in urine thromboxane between treatment groups
Urine 8 iso prostaglandin | 12 weeks
  Changes in urine 8 iso prostaglandin between treatment groups
Endothelial function by EndoPAT | 12 weeks
  Changes in endothelial function by EndoPAT (Endothelial Peripheral Arterial Tone) between treatment groups
Soluble markers of circulating adhesion molecules (VCAM, ICAM). | 12 weeks
  Changes in soluble markers of circulating adhesion molecules (VCAM, and ICAM) between treatment groups
hsCRP | 12 weeks
  Changes in hsCRP between treatment groups
Oxidized LDL | 12 weeks
  Changes in Oxidized LDL between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Bliden, BS, MBA, Study Director — Inova Health Care Services
Locations (1):
- Inova Heart and Vascular Institute, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.